CLINICAL TRIAL: NCT03390751
Title: Atropine Weight and Risk of Postoperative Confusion After Hip Fracture Surgery or Prosthetic Surgery of the Lower Limb, in the Elderly
Brief Title: Atropine Weight and Risk of Postoperative Confusion in the Elderly
Acronym: ATROPAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/17/0202; 2017-A01847-46 (Registry Identifier: ANSM Register)
Record Dates: First submitted 2017-11-16; First posted 2018-01-04 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Aging
Keywords: atropinic drugs; confusion; elderly patients
MeSH Terms: conditions — Confusion | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aged patients: Data collection of patients admitted to the orthopedic department of the University Hospital of Toulouse for surgical management of a fracture of the upper end of the femur in emergency or for the installation of a hip or knee prosthesis.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The collection of data will be done by interrogation of the patient and his family / entourage and rereading of medical records

SUMMARY:
The identification of a high atropine load of treatment received during hospitalization as a predictor of postoperative confusion could have various benefits:

* Pharmacoepidemiological: identify factors associated with postoperative confusion
* Clinics: by favoring treatments with a low atropine load during anesthesia, the management of patients hospitalized in orthopedics. Similarly, stopping or re-evaluating treatments with a high atropine weight for scheduled surgery is an easy step to take.
* Socio-economic: by reducing the costs related to the occurrence of a confusional syndrome (over-treatment, prolonged hospital stay, loss of autonomy, institutionalization of patients...).

In total, the present study would improve the daily management of hospitalized patients and the practices of clinicians, by offering a decision-making aid.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the orthopedic department for surgical management of a fracture of the upper end of the femur in emergency or for the installation of a hip or knee prosthesis
* Patient able to understand and respond to the protocol
* No opposition to the collection of data of the patient or his / her designee

Exclusion Criteria:

* Pre-existing confusion to surgery, detected by the CAM scale
* Serious or moderate head trauma less than three months old
* Removing / installing prosthesis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The recruitment of patients will be ensured from the consultation of anesthesia or the entry into hospitalization by the anesthesia team of the orthopedic surgery department of the Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Association between atropine load of medications on the risk of postoperative confusion | up to 7 days
  Occurrence of a postoperative confusion syndrome performed by Confusion Assessment Method (CAM) scale once a day. The CAM is a validated scale as a diagnostic scale for confusional syndrome at the patient's bedside with four parts : 1) confusion and fluctuation of symptoms, 2) inattention, 3) disorganization of thought, 4) disorder of consciousness.
Atropinic load of drugs | up to 7 days
  The DURAN scale is the most recent and most comprehensive atropine load evaluation scale. This scale classifies the evaluated drugs into three categories: no anticholinergic power (atropine weight = 0), low anticholinergic activity (atropine weight = 1), high atropinic power (atropine weight = 3). All drugs received by the patient during 7 days will be classified with the Duran scale.

SECONDARY OUTCOMES:
Duration of hospitalization | Up to discharge, an average of ten days
  Number of days of hospitalization (days) between surgery and discharge. Association between atropinic load of drugs and duration of hospitalization will be evaluated.
Autonomy | Month 3
  Description of autonomy of the patient at three months of surgery evaluated by the Activity Daily Living scale (ADL). The ADL scale evaluates activities of daily living: washing, dressing, going to the bathroom, ensuring transfers, continence and food. Each item is rated according to a level of dependence: independent (1 point), with assistance (0.5 points), unable to achieve (0 points). A total of 6 points indicates a total autonomy, and 0 a total dependency.
Cognitive dysfunction | baseline
  Appearance postoperative cognitive dysfunction by the Mini Mental State (MMS). the total score of MMS wil be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Minville, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Pierre-Paul-Riquet University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No